CLINICAL TRIAL: NCT00869609
Title: Evaluation of Group Lifestyle Balance Maintenance Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Trevor J. Orchard, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO08120047
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: Diabetes Prevention; CVD Risk Reduction; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLB Traditional Maintenance (TM) (Active Comparator): Group Lifestyle Balance (GLB) program Traditional Maintenance: After completion of the GLB 12 core sessions, participants who are randomly assigned to GLB program Traditional Maintenance (TM) will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions.
  Interventions: Behavioral: GLB Traditional Maintenance (TM)
- GLB-Carb-focused Maintenance (CF) (Active Comparator): Group Lifestyle Balance (GLB) program Carb-focused Maintenance: After completion of the GLB 12 core sessions, participants randomly assigned to GLB Carb-focused Maintenance (CF) will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information regarding healthy carbohydrate intake and hunger management.
  Interventions: Behavioral: GLB-Carb-focused Maintenance (CF)

INTERVENTIONS:
Behavioral: GLB Traditional Maintenance (TM) — After completion of the GLB 12 core sessions, participants will be randomly assigned to either Group Lifestyle Balance (GLB) program traditional maintenance or GLB Carb-focused maintenance. Participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information on healthy carbohydrate intake and hunger management.
  Arms: GLB Traditional Maintenance (TM)
Behavioral: GLB-Carb-focused Maintenance (CF) — After completion of the GLB 12 core sessions, participants will be randomly assigned to either Group Lifestyle Balance (GLB) program traditional maintenance or GLB Carb-focused maintenance. GLB-CF participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information on healthy carbohydrate intake and hunger management.
  Arms: GLB-Carb-focused Maintenance (CF)

SUMMARY:
Heart disease is a leading cause of death in people in the United States. It is a major problem for those with diabetes. Conditions called the metabolic syndrome and pre-diabetes increase risk for diabetes and heart disease. The metabolic syndrome is a group of disorders that occur at the same time. Overall, one in four American adults has the metabolic syndrome. It is more common in people over the age of 40. The metabolic syndrome includes: 1) large waist size, 2) high triglycerides, 3) low HDL cholesterol, 4) high blood pressure and 5) high fasting blood sugar. People with the metabolic syndrome have at least three of these five risk factors. Pre-diabetes is considered to be present in those with high fasting blood sugar levels below the diabetes range.

Research has shown that type 2 diabetes and the metabolic syndrome may be prevented or delayed by making lifestyle changes. It is not known what will most help people continue these healthy changes over time. The purpose of this study is to look at ways to help people continue the healthy lifestyle changes they have made while taking part in a diabetes prevention program called Group Lifestyle Balance (GLB).

DETAILED DESCRIPTION:
Objective: To determine the effectiveness of the Group Lifestyle Balance (GLB) program with an added maintenance component focusing on carbohydrate reduction and hunger management when compared to the GLB program with traditional maintenance.

Research Design and Methods: The original Diabetes Prevention Program intervention was modified from a 16 session individual intervention to a 12 session group-based program called Group Lifestyle Balance (GLB). The Diabetes Prevention Support Center (DPSC) has been created to oversee the implementation of diabetes prevention and CVD risk reduction in various community settings. GLB is a 12-session group based program that focuses on a low fat diet, weight loss and physical activity. This evidence-based intervention is directed at those with pre-diabetes and/or the metabolic syndrome. A monthly maintenance component will be added which provides support in assisting individuals who have completed the 12-session course in the maintenance of healthy lifestyle changes.

The efficacy (in terms of weight reduction) of an added maintenance component focusing on carbohydrate reduction and hunger management will be compared to traditional maintenance. Participants will be randomly assigned to either GLB traditional maintenance (GLB-TM) or GLB and carbohydrate reduced maintenance (GLB-CRM). There will be two groups of approximately 15 subjects in each intervention assignment, for a total of approximately 30 subjects per intervention group and approximately 60 subjects taking part overall. Efficacy in both groups will be assessed by pre and post-intervention measures of diet (weight loss) and physical activity (the keystones of the intervention), as well as the achievement of the two goals: a 7% weight loss by the end of 6 months and 150 minutes of physical activity per week. Secondary outcomes to be evaluated include the reduction of global CVD risk, as assessed by the Framingham Score, the presence of metabolic syndrome (NCEP ATP III), and a fall in blood sugar. Repeat measures will be obtained at six months and one year for further evaluation and comparison.

ELIGIBILITY:
Inclusion Criteria:

Non-diabetic patients with metabolic syndrome AND/OR pre-diabetes are eligible for this project based on the following criteria:

1. Metabolic Syndrome:

   Patients with BMI ≥ 25 kg/m2, with at least 3 of the following risk factors for metabolic syndrome:
   * Waist circumference (>40 inches men, >35 inches women)
   * Blood pressure ≥130 mmHg (systolic) or ≥85 mmHg (diastolic) OR history of diagnosed hypertension
   * Low HDL level (<40mg/dL men, <50 mg/dL women)
   * Elevated triglyceride level ≥150 mg/dL
   * Fasting glucose ≥100mg/dL and <126mg/dL
2. Pre-diabetes:

Patients with a BMI ≥25 kg/m2 and pre-diabetes (fasting glucose ≥100 mg/dL and <126mg/dL)

All measures should have been taken within one year of enrollment into the study. A permission for physical activity form must be signed by the participant's physician in order to take part in the study.

Exclusion Criteria:

* Previous diabetes or diabetes diagnosed as a result of the screening
* Age <18 years old
* Women who are currently (or within past 6-weeks) pregnant or lactating
* Any patient deemed by their physician not to be a candidate
* Any patient planning to leave the area before the end of the GILS
* Any patient who is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor J Orchard, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Diabetes Prevention Support Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Diabetes Prevention Support Center of the University of Pittsburgh — http://www.diabetesprevention.pitt.edu
- See also: Long-term Strategies for Diabetes Prevention: Evaluation of the Group Lifestyle Balance Post-Core Sessions Focusing on Carbohydrate and Hunger Management — http://www.omicsonline.org/longterm-strategies-for-diabetes-prevention-2155-6156.S2-006.php?aid=4819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The project was implemented in two settings: the first within an urban University campus and the second at a suburban YMCA. Recruitment commenced in May 2009 and was completed in July 2009.
Groups:
- GLB Traditional Maintenance (TM): Group Lifestyle Balance (GLB) program Traditional Maintenance. Participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions.
  GLB Traditional Maintenance: Group Lifestyle Balance (GLB)-Carb-focused Maintenance: Participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information on healthy carbohydrate intake and hunger management.
- GLB-Carb-focused Maintenance (CF): After completion of the GLB 12 core sessions, participants will be randomly assigned to either Group Lifestyle Balance (GLB) program traditional maintenance or GLB Carb-focused maintenance. GLB-CF participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information regarding healthy carbohydrate intake and hunger management.
  GLB-Carb-focused Maintenance: After completion of the GLB 12 core sessions, participants will be randomly assigned to either Group Lifestyle Balance (GLB) program traditional maintenance or GLB Carb-focused maintenance. GLB-CF participants will attend monthly maintenance sessions to assist them in maintaining the healthy lifestyle they have adopted during the 12 Core sessions. In addition, they will receive information on healthy carbohydrate intake and hunger management.
Period: Overall Study
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Started | 31 | 29
Completed | 25 | 26
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF) | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.4) | 53.4 (11.6) | 54.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Weight was measured twice without shoes with the average computed; participants were asked to remove their shoes at each measure.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Intention to treat analyses were performed; for those with missing weights at the post-intervention, 8 and 12 month visits, the last documented observation was carried forward. This information was available from the session data, where weight was collected weekly.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 31 | 29
pounds | 2.1 (5.9) | 0.2 (7.1)

2. Secondary Outcome: Change in Total Cholesterol
Description: Total cholesterol was measured after at least an eight-hour fast using the Cholestech LDX System by a certified research assistant.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with medication changes relevant to the outcome were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 28
mg/dl | 8.6 (23.2) | 15.4 (23.7)

3. Secondary Outcome: Change in HDL Cholesterol
Description: High-density lipoprotein (HDL) cholesterol was measured after at least an eight-hour fast using the Cholestech LDX System by a certified research assistant.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with medication changes relevant to the outcome were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 28
mg/dl | 2.9 (7.0) | 5.1 (6.4)

4. Secondary Outcome: Change in LDL Cholesterol
Description: Low-density lipoprotein (LDL) cholesterol was measured after at least an eight-hour fast using the Cholestech LDX System by a certified research assistant.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with medication changes relevant to the outcome were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 27
mg/dl | 5.2 (20.0) | 5.8 (23.3)

5. Secondary Outcome: Change in Triglycerides
Description: Triglycerides were measured after at least an eight-hour fast using the Cholestech LDX System by a certified research assistant.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 27
mg/dl | -0.003 (0.22) | -0.006 (39)

6. Secondary Outcome: Change in Fasting Glucose
Description: Fasting plasma glucose was measured after at least an eight-hour fast using the Cholestech LDX System by a certified research assistant.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 31 | 27
mg/dl | 1.2 (4.7) | 0.2 (6.9)

7. Secondary Outcome: Change in Glycosylated Hemoglobin A1c (HbA1c)
Description: Collected via venous blood draw, the HbA1c level reflects glucose concentration over the previous period (approximately 8-12 weeks, depending on the individual) and provides an indication of long-term glycemic control.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 31 | 28
percentage of glycosylated hemoglobin | -0.06 (0.18) | -0.08 (.18)

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: Blood pressure was measured in a sitting position in the right arm after resting for five minutes. First appearance and last heard (phase V) Korotkoff's sounds were used to define the pressure readings; the measures were repeated twice with a thirty second wait between each reading.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 24
mmHg | -0.43 (10.5) | -3.6 (10.8)

9. Secondary Outcome: Change in Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 27 | 24
mmHg | -2.1 (7.0) | -3.2 (8.8)

10. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference was measured at the midpoint between the lower rib margin and the iliac crest; the measurement was repeated twice and the average computed.
Time Frame: Measured at 8 months post intervention and 4 months post-randomization to maintenance group
Population: Participants with relevant medication changes were excluded.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Number analyzed (Participants) | 31 | 29
inches | -0.4 (1.3) | -0.2 (1.4)

ADVERSE EVENTS:
Time Frame: Approximately 1 year.
Arm/Group | GLB Traditional Maintenance (TM) | GLB-Carb-focused Maintenance (CF)
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

LIMITATIONS AND CAVEATS:
The sample size was small and included primarily white individuals, so these results may not be generalizable to other groups. The CPC was not carbohydrate restricted and may not be directly comparable to studies that focus on carbohydrate reduction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No